CLINICAL TRIAL: NCT05885243
Title: Evaluation of the Efficiency of ESWT and Custom İnsoles Produced With Podometric Measurement in the Treatment of Painful Heel Spurs
Brief Title: Evaluation of the Efficiency of ESWT and Custom İnsoles Produced With Podometric Measurement in the Treatment of Painful Heel Spurs (ESWT: Extracorporeal Shock Wave Therapy)
Acronym: eswt
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Bezmialem Vakif University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 4.2019/10
Record Dates: First submitted 2023-05-23; First posted 2023-06-01 (Actual); Last update posted 2023-06-01 (Actual); Status verified 2023-05

CONDITIONS: Heel Spur; Heel Spur Syndrome; Heel Pain Syndrome
Keywords: heel spur; extracorporeal shock wave therapy; insole; customized insole
MeSH Terms: conditions — Heel Spur; Fasciitis, Plantar

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- ESWT (Experimental): Group 1 (n:16) will be given once a week, total 5 sessions of ESWT+ home exercise program
  Interventions: Device: ESWT
- customized insoles (Experimental): Group 2 (n:16) will be given customized insoles+ home exercise program. Insoles will be used for 12 weeks.
  Interventions: Device: customized insoles
- combined ESWT and customized insoles (Experimental): Group 3 (n:16) will be given once a week, total 5 sessions of ESWT+ home exercise program. Also, simultaneous insoles will be provided. Insoles will be used for 12 weeks.
  Interventions: Device: ESWT; Device: customized insoles; Combination Product: combined ESWT and custtomized insoles

INTERVENTIONS:
Device: ESWT — will be given once a week, total 5 sessions ofESWT+ home exercises program
  Other Names: Home exercise program( strengthening, stretching exercises, frozen water bottle rolling)
  Arms: ESWT; combined ESWT and customized insoles
Device: customized insoles — Will be given customized insoles+ home exercise program. Insoles will be used for 12 weeks.
  Other Names: Home exercise program( strengthening, stretching exercises, frozen water bottle rolling)
  Arms: combined ESWT and customized insoles; customized insoles
Combination Product: combined ESWT and custtomized insoles — Will be given once a week, total 5 sessions of ESWT+ home exercise program. Also, simultaneous insoles will be provided. Insoles will be used for 12 weeks.
  Other Names: Home exercise program( strengthening, stretching exercises, frozen water bottle rolling)
  Arms: combined ESWT and customized insoles

SUMMARY:
The aim of the study; to determine the effectiveness customized insoles produced by podpmetric analysis and ESWT in patients with painfull heel spur and to determine the superiority of the treatments to each other.

DETAILED DESCRIPTION:
Heel spurs are the most common cause of heel pain in adults. Pain that occurs in heel spur and radiates to the soles of the feet is characteristic of this disease. The pain is most severe in the first steps after rest. Patients typically complain of severe pain on the first steps after getting out of bed in the morning. The pain is partially relieved after a few steps, but may increase again after intense activities. Typical pain history and examination findings are important to diagnose heel spur, and the diagnosis is confirmed by lateral x-ray. Generally, most patients with heel spurs benefit from conservative and medical treatment, and only a few need surgery. These treatment methods include many options such as activity and shoes modifications, topical and oral NSAIDs, insoles, stretching and strengthening exercises, various injections. TENS, ultrasound, electrotherapy modalities that can be used in therapy to relieve pain and promote healing.

Although many studies have been done for ESWT and insoles, there is not any study that comperes these two modalities. In this study, our aim is to investigate the effects of using ESWT and customized insoles alone or together on pain and foot functions in patients with heel spurs.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18-65 years
* Pain in the heel for at least 3 weeks
* Confirmation of the diagnosis with lateral foot radiography

Exclusion Criteria:

* Be younger than 18 and older than 65
* Patients with systemic rheumatological disease (rheumatoid arthritis, ankylosing spondylitis etc.)
* Entrapment neuropathy in the lower extremities
* Systemic active infection
* Malignancy
* Pregnancy
* Coagulopathy
* Patients who have had a previous heel injection of steroids
* Patients who received physical therapy from the heel area in the last 6 weeks (TENS, ultrasound, hotpack, etc.)
* Inserted cardiac pacemaker
* Underweight, obese, and morbidly obese according to BMI
* Patients using NSAIDs and myorelaxants continuously

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2023-06-15 (Estimated); Study Completion 2023-06-15 (Estimated)

PRIMARY OUTCOMES:
Visual Analog Scale | Change from baseline at 12 weeks after treatment.
  The self-evaluation of pain severity during rest, stretching and pressing on the medial calcaneal tubercle was calculated using a 10 cm VAS scale
American Orthopaedic Foot and Ankle Society (AOFAS) Pain Subscale | Change from baseline at 12 weeks after treatment.
  AOFAS scale includes three subscales (pain, function and alignment). Pain consists of one item with a maximal score of 40 points, indicating no pain.
Foot Function Index Pain Subscale | Change from baseline at 12 weeks after treatment.
  A Foot Function Index (FFI) was developed in 1991 to measure the impact of foot pathology on function in terms of pain, disability and activity restriction. The pain subcategory consists of 9 items and measures foot pain in different situations, such as walking barefoot versus walking with shoes.

SECONDARY OUTCOMES:
Roles and Maudsley Score | Change from baseline at 12 weeks after treatment.
  The Roles and Maudsley Score was used to evaluate pain and activity limitation as classified in four categories.1 point = excellent, 2 points = good, 3 points = fair and 4 points = poor
American Orthopaedic Foot and Ankle Society (AOFAS) Score | Change from baseline at 12 weeks after treatment.
  The AOFAS Ankle-Hindfoot Score is commonly used in patients with an ankle or hindfoot injury. This instrument combines functional outcome and pain, which are both critical for patients. The score consists of 3 subscales including alignment, pain, and function.
Foot Function Index | Change from baseline at 12 weeks after treatment.
  A Foot Function Index (FFI) was developed in 1991 to measure the impact of foot pathology on function in terms of pain, disability and activity restriction.

CONTACTS AND LOCATIONS:
Overall Officials: Okan Küçükakkaş, Doç, Study Director — okan4494@yahoo.com; Nesrin Yılmaz Baıramov, MD, Principal Investigator — nsrn.ylmz@yahoo.com; Elif Uğurlu, MD, Study Chair — elifdemirbag92@gmail.com
Locations (1):
- Bezmialem Vakif University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wrobel JS, Fleischer AE, Crews RT, Jarrett B, Najafi B. A randomized controlled trial of custom foot orthoses for the treatment of plantar heel pain. J Am Podiatr Med Assoc. 2015 Jul;105(4):281-94. doi: 10.7547/13-122.1. Epub 2015 May 5. PMID 25941995
- [Background] Yan W, Sun S, Li X. [Therapeutic effect of extracorporeal shock wave combined with orthopaedic insole on plantar fasciitis]. Zhong Nan Da Xue Xue Bao Yi Xue Ban. 2014 Dec;39(12):1326-30. doi: 10.11817/j.issn.1672-7347.2014.12.017. Chinese. PMID 25544167
- [Background] Cohena-Jimenez M, Pabon-Carrasco M, Perez Belloso AJ. Comparison between customised foot orthoses and insole combined with the use of extracorporeal shock wave therapy in plantar fasciitis, medium-term follow-up results: A randomised controlled trial. Clin Rehabil. 2021 May;35(5):740-749. doi: 10.1177/0269215520976619. Epub 2020 Nov 24. PMID 33233945
- [Background] Caglar Okur S, Aydin A. Comparison of extracorporeal shock wave therapy with custom foot orthotics in plantar fasciitis treatment: A prospective randomized one-year follow-up study. J Musculoskelet Neuronal Interact. 2019 Jun 1;19(2):178-186. PMID 31186388
- [Background] Ribeiro AP, de Souza BL, Joao SMA. Effectiveness of mechanical treatment with customized insole and minimalist flexible footwear for women with calcaneal spur: randomized controlled trial. BMC Musculoskelet Disord. 2022 Aug 13;23(1):773. doi: 10.1186/s12891-022-05729-4. PMID 35964021
- [Background] Landorf KB, Keenan AM, Herbert RD. Effectiveness of foot orthoses to treat plantar fasciitis: a randomized trial. Arch Intern Med. 2006 Jun 26;166(12):1305-10. doi: 10.1001/archinte.166.12.1305. PMID 16801514